CLINICAL TRIAL: NCT07303322
Title: Phase 3, Prospective, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Clinical Trial to Evaluate the Efficacy and Safety of N1087 in Participants With Female Pattern Hair Loss
Brief Title: Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of N1087 in Participants With Female Pattern Hair Loss (MINORA-WOMEN)
Acronym: MINORA-WOMEN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EF193A
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Female Pattern Hair Loss; Female Pattern Hair Loss, Androgenic Alopecia
Keywords: Androgenetic Alopecia; Hair Loss; Female Pattern Hair Loss; Alopecia; Randomized Controlled Trial; Phase 3
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 2:1 to receive N1087 or placebo. The intervention includes an 8-week dose titration (0.5 mg, 1 mg, 1.5 mg, 2 mg, each for 2 weeks), followed by 16 weeks at the maximum tolerated dose (up to 2 mg/day). Randomization will be stratified by Sinclair scale (2-4) and age (<40 or ≥40). Multicenter, Brazil.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N1087 (Experimental): Participants will receive N1087, starting at 0.5 mg/day and titrated every 2 weeks (1 mg, 1.5 mg, up to 2 mg/day) during an 8-week titration period, followed by 16 weeks at the maximum tolerated dose (up to 2 mg/day). Administered orally once daily for a total of 24 weeks.
  Interventions: Drug: N1087
- Placebo (Placebo Comparator): Participants will receive placebo, administered once daily for 24 weeks, following the same titration schedule as the experimental arm to maintain blinding.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N1087 — N1087 is an oral solution administered in drops. Treatment begins with an 8-week titration period: 0.5 mg/day for 2 weeks, then 1 mg/day, 1.5 mg/day, and up to 2 mg/day every 2 weeks. After titration, participants continue for 16 weeks at the maximum tolerated dose (up to 2 mg/day). Administered orally once daily for a total of 24 weeks.
  Arms: N1087
Drug: Placebo — Placebo administered once daily for 24 weeks, following the same titration schedule as the experimental arm to maintain blinding.
  Arms: Placebo

SUMMARY:
This is a Phase 3, prospective, randomized, double-blind, placebo-controlled, parallel-group, multicenter clinical trial designed to evaluate the efficacy and safety of N1087 in women with female pattern hair loss (FPHL). Participants will receive either N1087 or placebo for 24 weeks. The study includes a titration period starting at 0.5 mg and increasing up to 2 mg daily, followed by treatment at the maximum tolerated dose. The primary objective is to assess changes in non-vellus hair density in the target scalp area after 24 weeks. Secondary objectives include changes in terminal hair density, hair thickness, global photographic assessment, quality of life, and participant satisfaction. Safety will be monitored through adverse events, vital signs, and laboratory tests. Approximately 372 participants will be randomized in a 2:1 ratio (N1087 vs. placebo) across about 10 research centers in Brazil.

DETAILED DESCRIPTION:
This Phase 3 clinical trial is a prospective, randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate the efficacy and safety of N1087 in women with female pattern hair loss (FPHL), also known as female androgenetic alopecia. FPHL is a chronic, progressive condition characterized by gradual thinning of hair and reduced density, primarily in the frontal and vertex regions of the scalp. Current treatment options are limited, and topical minoxidil, although widely used, is not approved for women in Brazil and presents adherence challenges. Low-dose oral minoxidil has shown promising efficacy and safety in clinical practice and literature, but high-quality controlled trials are lacking.

Participants will be randomized in a 2:1 ratio to receive N1087 or placebo for 24 weeks. The intervention begins with an 8-week titration period (0.5 mg/day for 2 weeks, then 1 mg, 1.5 mg, and 2 mg every 2 weeks) followed by 16 weeks at the maximum tolerated dose (up to 2 mg/day). The primary endpoint is the change from baseline in non-vellus hair density (≥0.03 mm diameter) in the target area at Week 24, assessed by standardized digital phototrichogram. Secondary endpoints include changes in terminal hair density, total hair density, hair shaft thickness, reversal of follicular miniaturization, global photographic assessment (Investigator Global Assessment), quality of life (WAA-QoL questionnaire), and participant satisfaction. Safety assessments include adverse events, vital signs, ECG, and laboratory tests.

The study will enroll approximately 372 participants across 10 sites in Brazil, with eligibility criteria including women aged 18-60 years, Sinclair scale 2-4, and no recent treatments for FPHL. Exclusion criteria include other causes of alopecia, uncontrolled hypertension, cardiovascular conditions, hormonal disorders, and pregnancy. The total study duration per participant is approximately 36 weeks (up to 12 weeks screening/washout, 8 weeks titration, 16 weeks treatment). A Data Monitoring Committee will oversee safety.

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged ≥18 years and ≤60 years at the time of signing the informed consent form.
* Presentation of female pattern hair loss in stages 2 to 4 of the Sinclair scale (Women's Alopecia Severity Scale - WASS), based on the Investigator's clinical examination.
* Absence of specific treatment for female pattern hair loss (FPHL) in the last 6 months or history of specific treatment for FPHL lasting ≤30 days in the last 6 months. Participants currently using specific treatment for FPHL or with prior use lasting >30 days in the last 6 months must complete a 3-month washout period before the Randomization Visit (RV).
* Willing to agree to all procedures and assessments required by the clinical trial, including a permanent tattoo applied to the scalp and shaving of the target area.
* Willing to maintain hair style, length, and color throughout the study.
* Willing to maintain consistent use of hair care products and general hair care routine during the entire study.

Exclusion Criteria:

* Participant presenting other causes of alopecia, such as: alopecia areata, scarring alopecia, traction alopecia, nutritional deficiency, monilethrix, trichotillomania, trichothiodystrophy, chemotherapy-induced alopecia.
* Participant who experienced telogen effluvium in the last 6 months, such as after childbirth, infection, intense stress.
* Participant presenting other dermatological conditions on the scalp, such as: seborrheic dermatitis, psoriasis, eczema, scalp mycosis.
* Participant presenting signs or symptoms of hyperandrogenism, such as: hirsutism, moderate to severe acne.
* Participant with previous diagnosis of hormonal disorders, such as: polycystic ovary syndrome, ovarian or adrenal tumors.
* Participant with previous diagnosis of pituitary disorders, such as: prolactinoma, panhypopituitarism.
* Participant presenting uncontrolled thyroid disease.
* Participant with previous diagnosis of autoimmune diseases or collagen disorders, such as: systemic lupus erythematosus, dermatomyositis, scleroderma.
* Participant in use of hormonal therapy initiated or changed in the last 6 months.
* Participant who has received an organ transplant.
* Participant who underwent physical treatments for hair loss in the last 6 months, such as: microneedling, laser, platelet-rich plasma. Note: in this case, the participant must complete a 3-month washout period.
* Participant with history of hair transplant.
* Participant who uses hair extensions.
* Participant presenting severe uncontrolled hypertension (systolic blood pressure [SBP] >180 mmHg or diastolic blood pressure [DBP] >110 mmHg).
* Participant presenting confirmed orthostatic hypotension (sustained reduction of SBP ≥20 mmHg or DBP ≥10 mmHg within 3 minutes after standing).
* Participant presenting arterial hypotension (SBP <90 mmHg or DBP <60 mmHg).
* Participant with previous diagnosis or suspected pulmonary hypertension associated with mitral stenosis.
* Participant with previous diagnosis of acute myocardial infarction.
* Participant with previous diagnosis or suspected pheochromocytoma.
* Participant presenting history of peripheral edema, lymphedema, or ascites.
* Participant with history or risk factor for pericardial effusion.
* Participant with previous diagnosis of other moderate to severe cardiovascular, renal, or hepatic diseases.
* History of any malignancy in the last 5 years, except successfully treated non-metastatic basal cell or squamous cell carcinoma of the skin.
* Participant in current use of potent vasodilators, such as: hydralazine and isosorbide.
* Participant with known allergy or hypersensitivity to minoxidil or any component of the formulation.
* Participant presenting hair styles that, in the Investigator's opinion, prevent study assessments, such as: permanent braids, dreadlocks, box braids, nagô.
* Participant who is pregnant, breastfeeding, or has potential to become pregnant and does not agree to use a contraceptive method during the clinical trial.
* Participant presenting any clinically significant condition that, in the Investigator's opinion, makes the participant unsuitable for participation in the trial.
* Participant who has participated in clinical trial protocols in the last 12 months, unless the Investigator considers there may be direct benefit.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372 (Estimated)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in non-vellus hair density (≥0.03 mm diameter) in the target scalp area at Week 24 | 24 weeks
  Non-vellus hair density (≥0.03 mm diameter) will be measured in the target scalp area using standardized digital phototrichogram. The primary endpoint is the absolute change from baseline to Week 24.